CLINICAL TRIAL: NCT04105465
Title: Randomised,Crossover, Feasibility Study to Evaluate the PlasmaJet in the Management of Lymphedema and Lymphocyst Formation in Patients Undergoing Bilateral Groin Node Dissection (BGND) for Vulval Cancer
Brief Title: Study to Evaluate the Role of PlasmaJet in Patients Undergoing Groin Node Dissection for Vulval Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Conflict with another study that was opened to recruitment
Sponsor: Royal Surrey County Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Thumuluru Kavitha Madhuri, Senior Clinical Fellow, Royal Surrey County Hospital NHS Foundation Trust
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PJBGNDRSCH
Record Dates: First submitted 2019-02-11; First posted 2019-09-26 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Vulvar Cancer; Groin Node
Keywords: vulvar cancer; groin node dissection; bilateral groin node dissection; lymphedema; lymphocyst; lymphorrea
MeSH Terms: conditions — Vulvar Neoplasms; Lymphedema; Lymphocele

STUDY DESIGN:
Intervention Model Description: The trial design was conceived as a single site, double blind, crossover study in which each patient would be their own control would offer the most useful information.
Who Masked: Participant, Outcomes Assessor
Masking Description: A double blind system was applied. Since randomisation was performed in theatre, the patient was unaware of the side that the PJ device was applied. This was not mentioned in the operation notes either. As a result, the nursing team on the inpatient ward were also blinded to the randomisation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Surgery without trial (PJ) device (No Intervention): All steps of surgery are conducted as per standard practice in accordance with the current practice at the time. In all cases a bilateral inguino-femoral groin node dissection was performed, with en-bloc removal of the superficial and deep inguinal nodes with conservation of the long saphenous vein.
- Surgery with trial (PJ) device (Active Comparator): Use of the PJ was limited to the randomised side only. All steps of surgery are conducted as per standard practice in accordance with the current practice at the time. In all cases a bilateral inguino-femoral groin node dissection was performed, with en-bloc removal of the superficial and deep inguinal nodes with conservation of the long saphenous vein. Haemostasis was ensured with diathermy and ties and just prior to wound closure, the surgeon used the PlasmaJet on the indicated groin to seal the lymph vessels and channels at a setting of 40% by spraying the argon plasma over the entire exposed surgical field at a distance of 10 mm from the surface to the tip of the instrument.
  Interventions: Device: PlasmaJet

INTERVENTIONS:
Device: PlasmaJet — The PlasmaJet device is used following groin node dissection on the side randomised to receive it as per protocol specifications
  Arms: Surgery with trial (PJ) device

SUMMARY:
Surgery for vulvar cancer involves removal of the central tumour as well as groin node dissection as indicated depending on the stage of tumour. Groin node dissection is associated with significant complications including lymphorrea, lymphocyst formation, wound breakdown as well as long term complications including lymphedema.

This study has been designed with each patient acting as their own control to investigate if using the PlasmaJet during surgery is associated with a reduction in the above mentioned complications.

DETAILED DESCRIPTION:
Vulvar malignancy is the fourth most common malignancy of the female genital tract. Surgical excision achieves excellent local control and remains the mainstay of treatment.

Surgical excision depends on the extent of disease and may be in the form of wide local excision or radical vulvectomy. Lymphadenectomy in the form of bilateral groin node dissection (BGND) is performed for all central tumors with depth of invasion greater than 1 mm, unless there is significant comorbidity contraindicating this, but is known to cause significant postoperative morbidity. Immediate postoperative complications include breakdown and lymphocyst formation in more than 50% of cases. The PlasmaJet is a novel device that produces a jet of pure argon plasma by heating pressurized argon gas. Energy from the argon plasma transfers to tissue as light, heat, and kinetic energy.

Following ethical approval, a prospective, crossover, doubleblind, randomized, control trial to assess the PJ system, with the primary outcome being the possibility of reduction in wound breakdown and lymphocyst and lymphedema formation following BGND for vulvar cancer was opened.

ELIGIBILITY:
Inclusion Criteria:

* To be included in this study, all women should undergo BGND during their treatment pathway for histologically confirmed vulval cancer.
* Participant is willing and able to provide informed consent.
* Aged 18 years or above.
* Participant willing to allow General Practitioner and other health care professionals, if appropriate, to be notified of participation in study.

Exclusion Criteria:

* Women with vulval cancer who do not undergo BGND.
* Women with any previous groin surgery
* Women with any previous radiotherapy to the pelvic area including the groins
* Patient choice
* Women who are pregnant, lactating or planning pregnancy during the course of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women undergoing BGND during their treatment pathway for histologically confirmed vulval cancer
Enrollment: 21 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment into the pilot study.The rate (% and absolute rate) of recruitment | 24 months

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | Upto 1 year following surgery
  To document the side-effect profile post-operatively following surgery with the PJ device.
Risk of groin lymphorrea/ lymphocyst formation using daily drain outputs | Upto 1 year following surgery
  To explore the potential and safety of the PJ device in the prevention of groin lymphocyst formation by prophylactic coagulation of lymph vessels in patients undergoing BGND for vulval cancer
Wound Infection | Upto 3months following surgery or till groins healed whichever is sooner
  Rate of wound infection following standard surgery vs PlasmaJet use in the groins will be assessed
Length of Stay | Until 14 days following surgery
  Length of hospital stay following surgery will be recorded as well as any readmissions
Lymphedema using the CTC V3.0 grading system | Upto two years following study entry
  Grade of lymphedema to be assessed at each clinic visit for two years following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Thumuluru K Madhuri, MD, Principal Investigator — Royal Surrey County Hospitals NHS Foundation Trust
Locations (1):
- Department of Gynaecological Oncology, Royal Surrey County Hospital NHS Foundation Trust, Guildford, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No patient indentifiable data will be shared however anonymised data can be made available on request